CLINICAL TRIAL: NCT02917057
Title: A Cohort Study of the Benefits of Bydureon in Customary Clinical Care in the United States - Additional Analyses
Brief Title: Subanalyses of Elderly Type 2 Diabetes Patients or Type 2 Diabetes Patients With Renal Impairment
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5551R00011
Record Dates: First submitted 2016-09-08; First posted 2016-09-28 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exenatide once weekly initiators: Type 2 diabetes patients who initiated exenatide once weekly treatment during the index period
  Interventions: Drug: exenatide once weekly
- Basal Insulin initiator cohort: Type 2 diabetes patients who initiated basal insulin treatment in the index period
  Interventions: Drug: basal insulin

INTERVENTIONS:
Drug: exenatide once weekly — Exenatide treatment in customary clinical care in the USA
  Groups: Exenatide once weekly initiators
Drug: basal insulin — basal insulin tretament in the customary clinical care in USA
  Groups: Basal Insulin initiator cohort

SUMMARY:
Exenatide once weekly (Bydureon) was approved in January 2012 by FDA in USA for the treatment of type 2 diabetes mellitus. Evidence from clinical trials suggested that Bydureon improves glucose control with low risk of hypoglycemia. Bydureon does not require a dose titration as necessary for other glucagon-like peptide-1 agonists, and appears to have other advantages, such as reducing insulin resistance, reducing weight, and improving blood pressure and lipid profiles. However, the degree to which these advantages of Bydureon lead to improve outcomes in customary clinical care in patients with mild and moderate renal impairment and in elderly patients are unknown.

The aim of this study is to evaluate the effectiveness and tolerability of Bydureon relative to basal insulin initiated as first-ever injectable therapeutic regimens among elderly patients and patients with renal impairment. Patients who initiated treatment with Bydureon or basal insulin between July 2011 and March 2015 will be recruited into the study cohorts from Optum's database of electronic health records. The two treatment cohorts will be matched by propensity score method. Changes in HbA1c, weight, markers for renal function (estimated glomerular filtration rate (eGFR), serum creatinine, and albumin/creatinine ratio (ACR)), and incidences of gastrointestinal symptoms and hypoglycaemia are investigated for patients with different eGFR categories and with different ages.

DETAILED DESCRIPTION:
Background: In January 2012, the US Food and Drug Administration approved a once-weekly form of exenatide, Bydureon, for the treatment of type 2 diabetes mellitus. Evidence from clinical trials suggested that Bydureon improves glucose control with low risk of hypoglycemia. Bydureon does not require a dose titration as necessary for other glucagon-like peptide-1 agonists (GLP-1RAs), and appears to have other advantages, such as reducing insulin resistance, reducing weight, and improving blood pressure and lipid profiles. However, the degree to which these advantages of Bydureon lead to improve outcomes in patients with renal impairment or who are elderly is unknown.

Aims: The aim of this study is to evaluate the effectiveness and tolerability of Bydureon relative to basal insulin initiated as first-ever injectable therapeutic regimens among elderly patients and patients with renal impairment.

The specific study objectives are as follows:

* To quantify the effectiveness of Bydureon initiation relative to initiation of basal insulin, on improving:
* Glycated hemoglobin (HbA1c)
* Weight (body mass index (BMI))
* HbA1c simultaneous to reduction in weight
* Blood pressure and lipid profiles
* To examine the tolerability of Bydureon initiation relative to initiation basal insulin, on the occurrence of :
* Hypoglycemia
* Gastrointestinal symptoms (nausea, vomiting, diarrhea, and constipation)
* Change in the markers for renal function (estimated glomerular filtration rate (eGFR), serum creatinine, and albumin/creatinine ratio (ACR), and the stability of liver function test (AST, ALT) and standard blood counts (WBC, RBC, HCT, Hgb, PLT)
* To examine these measures of effectiveness and tolerability within potentially vulnerable subgroups of Bydureon and basal insulin initiators:
* T2D patients with renal impairment
* Elderly T2D patients Study Population and Design: This retrospective cohort study will use Optum's EHR data from July 2011 through March 2015 and identify injectable-naive T2D patients who initiated either Bydureon or basal insulin during the accrual period, January 2012 and January 2015. Injectable-naive T2D patients will be indetified. Propensity score methods will be used to match Bydureon initiators with basal insulin initiators.

Subgroup Comparisons: Within the EHR data, serum creatinine values will be used to calculate the eGFR using an equation developed by the Chronic Kidney Disease (CKD) Epidemiology (EPI) Collaboration, called the CKD-EPI Equation.

Renal Impairment: Patients will be stratified by eGFR ranges in baseline indicative of the renal impairment, as follows:

* Normal, eGFR ≥ 90.00 mL/min/1.73m2
* Mild impairment, 60.00 < eGFR < 89.99 mL/min/1.73m2
* Moderate and Severe impairment, eGFR < 59.99 mL/min/1.73m2

Elderly T2D Patients: Elderly subgroups will be defined as 65+ years of age. Patients will be stratified by age on index date, as follows:

* < 65 years
* 65 to 74 years
* 75+ years Outcomes and Analysis: To measure the effectiveness of Bydureon relative to basal insulin are changes in HbA1c and body weight, as well as changes in HbA1c and simultaneous reduction in weight. Changes in BMI, lipid profiles, and blood pressure will be assessed. These variables are part of the clinical and laboratory data in the EHR. Each outcome will be evaluated for completeness, multiply imputed, and reported across standardized time intervals. HbA1c, weight and BMI will be summarized in baseline and quarterly (3-month intervals) in the first year following drug initiation. Lipid measurements and blood pressure will be summarized in baseline and bi-annually (6-month intervals) in the first year following drug initiation.

To assess drug tolerability, incidence of hypoglycemia, and gastrointestinal symptoms (nausea, vomiting, diarrhea, and constipation) will be calculated. These outcomes will be ascertained using an ICD-9 algorithm applied to the structured fields and by extracting mentions of hypoglycemia using a natural language processing (NLP) algorithm developed by Optum and applied to the free text clinical notes available in the data. In addition the stability of renal function evaluated by change in eGFR, or albumin/creatinine ratio (ACR); the change in serum hepatic enzymes [aspartate aminotransferase (AST), alanine aminotransferase (ALT)], and hematologic measures [red blood cells counts (RBC), white blood cell counts (WBC), platelets (PLT), hemoglobin (Hgb) and hematocrit (Hct) will be evaluated. Each of these laboratory values will be evaluated for completeness, multiply imputed, and reported across standardized time intervals. eGFR and ACR are summarized in baseline and quarterly (3-month intervals) in the first year following drug initiation. Hepatic enzymes and hematologic measures are summarized in baseline and semi-annually (6-month intervals) in the first year following drug initiation.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old;
* had received care documented in EHR (including at least one out-patient provider visit) for a minimum of 6-months prior index date;
* had at least one diagnosis of Type 2 diabetes (ICD-9-CM: 250.X0 or 250.X2) prior to and including the date of the study drug initiation, with no prior diagnosis of type1 diabetes (ICD-9-CM: 250.X1 or 250.X3), or gestational diabetes within the 6-months prior to index date;
* No evidence of prior injectable antidiabetic treatment, specifically no dispensing of a GLP-1-RA or any insulin during the 6-months baseline period prior to study drug initiation

Exclusion Criteria:

* Prior diagnosis of type 1 diabetes (ICD-9-CM: 250.X1 or 250.X3), or gestational diabetes within the 6-months prior to index date;
* Prior dispensing of a GLP-1RA or any insulin
* Missing data on renal function defined by eGFR or age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population was drawn from an Optum's Electronic Health Records (EHR) database. Injectable-naive type 2 diabetic patients who initiated therapy with either Exenatide once-weekly or basal insulin from January 2012 to January 2015, with follow-up through March 2015 were identified. The baseline period was defined as the 183 days (6-months) prior to date of study drug initiation (index date). Patients with Type 2 diabetes were identified using structured diagnosis fields and International Classification of Disease, Ninth Revision, Clinical Modification (ICD-9-CM) codes. Initiations of Exenatide once-weekly or basal insulin were identified in the EHR data capturing prescribed medications using National Drug Codes (NDC).
Sampling Method: Non-Probability Sample
Enrollment: 6024 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2015-08-01 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in HbA1c (%) | one year post-index
  To evaluate changes in HbA1c (%) from baseline after initiation of therapy with exenatide once-weekly in patients with different renal functions or age classes, as referred to basal insulin initiators of the same subgroups.
Changes from baseline in weight (kg) | one year post-index
  To evaluate changes in weight (kg) from baseline after initiation of therapy with exenatide once-weekly in patients with different renal functions or age classes, as referred to basal insulin initiators of the same subgroups.

SECONDARY OUTCOMES:
Changes from baseline in eGFR | one year post-index
  Changes in eGFR after initiation of therapy with exenatide once-weekly in patients with different renal functions or age classes, as referred to basal insulin initiators of the same subgroups.
Frequency of Hypoglycemia | one year post-index
  Frequency of episodes of hypoglycaemia after initiation of therapy with exenatide once-weekly in patients with different renal functions or age classes, as referred to basal insulin initiators of the same subgroups.
Frequency of Nausea | one year post-index
  Frequency of episodes of nausea after initiation of therapy with exenatide once-weekly in patients with different renal functions or age classes, as referred to basal insulin initiators of the same subgroups.
Frequency of Vomiting | one year post-index
  Frequency of episodes of vomiting after initiation of therapy with exenatide once-weekly in patients with different renal functions or age classes, as referred to basal insulin initiators of the same subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Anita M Loughlin, Ph.D, Principal Investigator — Optum, Inc.
Locations (1):
- Optum Epidemiology, Boston, Massachusetts, United States

REFERENCES:
- [Background] Loughlin AM, Qiao Q, Nunes AP, Ohman P, Ezzy S, Yochum L, Clifford CR, Gately R, Dore DD, Seeger JD. Effectiveness and tolerability of therapy with exenatide once weekly vs basal insulin among injectable-drug-naive elderly or renal impaired patients with type 2 diabetes in the United States. Diabetes Obes Metab. 2018 Apr;20(4):898-909. doi: 10.1111/dom.13175. Epub 2018 Jan 3. PMID 29193561
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4434&filename=D5551R00011_Poster_ADA2016.pdf